CLINICAL TRIAL: NCT01763567
Title: A Multi-Phased, Multi-Center Study to Evaluate Safety and Device Performance of the Medtronic Hospital Glucose Management System (HGMS) in Critically Ill Adult Patients
Brief Title: Feasibility Study to Evaluate Safety and Device Performance of the Hospital Glucose Management System (HGMS)
Acronym: MAHI
Status: Completed | Type: Observational
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Other Study IDs: CEP244
Record Dates: First submitted 2012-12-21; First posted 2013-01-09 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Hyperglycemia
Keywords: Medtronic; Diabetes; Hospital; Continuous Glucose Monitor; Intensive Care Unit
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess safety and device performance of the Medtronic Hospital Glucose Management System (HGMS) for up to 72-hours.

DETAILED DESCRIPTION:
Assess safety and device performance of the Medtronic HGMS in the critically-ill setting and analyze the following:

1. Device Performance:

   * Functionality of HGMS
   * Alerts/Alarms Specificity and Sensitivity
   * System Workflow
2. Safety:

   * Descriptive statistics will be used to characterize safety events
   * Moderate and severe anticipated device and procedure related adverse events
   * All serious adverse events and unanticipated adverse device effects related events

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old
2. Subject is admitted to the ICU
3. Subject has a treatment regimen that includes a glucose target range of ≥140 mg/dl
4. Subject has a treatment regimen that includes an intended continuous intravenous insulin for at least 24 hours

   a. Including patients with no previous diagnosis of Diabetes Mellitus
5. Subject has anticipated life expectancy greater than 96 hours
6. Subject has recent platelet count greater than 30,000 per micro-liter

Exclusion Criteria:

1. Subject currently has a suspected or diagnosed medical condition that, in the opinion of the Investigator, warrants exclusion from the study or prevents the subject from completing the study
2. Subject is currently participating in another investigational drug or device study
3. Subject is pregnant, as determined by hospital admission
4. Subject is receiving treatment that includes Hydroxyurea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit (ICU) and on intravenous (IV) insulin therapy for the treatment of transient or diabetes-related hyperglycemia
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Kosiborod, M.D, Principal Investigator — St Luke's Hospital - Mid America Heart Institute
Locations (1):
- St Luke's Hospital Mid America Heart Institute, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Kosiborod M, Gottlieb RK, Sekella JA, Peterman D, Grodzinsky A, Kennedy P, Borkon MA. Performance of the Medtronic Sentrino continuous glucose management (CGM) system in the cardiac intensive care unit. BMJ Open Diabetes Res Care. 2014 Jul 21;2(1):e000037. doi: 10.1136/bmjdrc-2014-000037. eCollection 2014. PMID 25452874

RESULTS

PARTICIPANT FLOW:
Groups:
- Oberservation Arm: To assess safety and device performance for the Hospital Glucose Managment system
Period: Overall Study
Arm/Group | Oberservation Arm
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Oberservation Arm
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Device Performance: Accuracy of HGMS
Description: Mean Absolute Relative Difference (MARD), calculated as the absolute difference of [(sensor glucose values - iSTAT glucose values) / iSTAT glucose values].
  The portable i-STAT handheld makes patient-side testing easy:
  * Requires no special sample preparation or user calibration; maintenance is minimal
  * Weighs 18 ounces, making it portable
  * Patient-side testing is as easy as entering the operator and patient information into the handheld, inserting one of the several filled test cartridges, and then viewing test results:
  * The system prompts users step by step through the testing process
  * Operator and patient information can be entered via barcode scanner
  * Operator lockout prevents unauthorized users from performing or viewing test results
  * Test results are uploaded automatically when the i-STAT handheld is placed in a downloader
Time Frame: up to 72 hours
Population: To assess safety and device performance for the Hospital Glucose Managment system
Measure: Mean (Standard Deviation); unit: percent difference
Arm/Group | Oberservation Arm
Number analyzed (Participants) | 19
percent difference | 12.8 (9.5)
Statistical Analysis 1: Comparison: Oberservation Arm; Test type: Superiority or Other; Mean Difference (Final Values) = 12.8, Standard Deviation 9.5

2. Other Pre Specified Outcome: Functionality of HGMS: Alerts and Alarms - % of Hypo Events Correctly Detected
Description: The device alarmed within 30 minutes before or after the reference blood glucose value (i-STAT) goes below 70 mg/dL setting levels. The % of hypo events correctly detected was calculated as: total number of correct events divided by total number of events from all 19 participants.
Time Frame: up to 72 hours
Measure: Number; unit: percentage of total events
Arm/Group | Oberservation Arm
Number analyzed (Participants) | 19
percentage of total events | 16.7
Statistical Analysis 1: Comparison: Oberservation Arm; Test type: Superiority or Other; percent of events correctly detected = 16.7

3. Other Pre Specified Outcome: Functionality of HGMS: Alerts and Alarms - % of Hyper Events Correctly Detected
Description: The device alarmed within 30 minutes before or after the reference blood glucose value (i-STAT) goes above 250 mg/dL setting levels. The % of hyper events correctly detected was calculated as: total number of correct events divided by total number of events from all 19 participants.
Time Frame: 72 hours
Measure: Number; unit: percentage of total events
Arm/Group | Oberservation Arm
Number analyzed (Participants) | 19
percentage of total events | 88.9
Statistical Analysis 1: Comparison: Oberservation Arm; Test type: Superiority or Other; percent of events correctly detected = 88.9

4. Other Pre Specified Outcome: Functionality of HGMS: Alerts and Alarms - % of Hypo False Alert
Description: Definition of % of hypo false alert: within 30 minutes before or after the sensor alarmed at 70 mg/dL, there is no reference blood glucose value (i-STAT) that goes below 70 mg/dL. The % of hypo false alert was calculated as: total number of false events divided by total number of events from all 19 participants. NOTE: % of Hypo False Alert and % Hypo Event Correctly Detected do not necessarily add up to 100% because the denomintors are not the same.
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of all alerts
Arm/Group | Oberservation Arm
Number analyzed (Participants) | 19
percentage of all alerts | 85.8
Statistical Analysis 1: Comparison: Oberservation Arm; Test type: Superiority or Other; % of false alert = 85.8

5. Other Pre Specified Outcome: Functionality of HGMS: Alerts and Alarms - % of Hyper False Alert
Description: Definition of % of Hyper False Alert: within 30 minutes before or after the sensor alarmed at 250 mg/dL, there is no reference blood glucose value (i-STAT) that goes above 250mg/dL . The % of hyper false alert was calculated as: total number of false events divided by total number of events from all 19 participants. NOTE: % of Hyper False Alert and % Hyper Event Correctly Detected do not necessarily add up to 100% because the denomintors are not the same.
Time Frame: Up to 72 hours
Measure: Number; unit: percentage of all alerts
Arm/Group | Oberservation Arm
Number analyzed (Participants) | 19
percentage of all alerts | 56.5
Statistical Analysis 1: Comparison: Oberservation Arm; Test type: Superiority or Other; % of false alert = 56.5

ADVERSE EVENTS:
Time Frame: 3 days for each subject
Groups:
- Observation Arm: To assess safety and device performance for the Hospital Glucose Managment system
Arm/Group | Observation Arm
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No